CLINICAL TRIAL: NCT04139317
Title: A Randomized, Open Label, Multicenter Phase II Study Evaluating the Efficacy and Safety of Capmatinib (INC280) Plus Pembrolizumab Versus Pembrolizumab Alone as First Line Treatment for Locally Advanced or Metastatic Non-small Cell Lung Cancer With PD-L1≥ 50%
Brief Title: Safety and Efficacy of Capmatinib (INC280) Plus Pembrolizumab vs Pembrolizumab Alone in NSCLC With PD-L1≥ 50%
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to terminate due to the lack of tolerability observed in patients treated with capmatinib and pembrolizumab in the combination arm as compared to patients treated with pembrolizumab alone in the pembrolizumab single agent arm
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CINC280I12201; 2019-002660-27 (EudraCT Number)
Record Dates: First submitted 2019-10-14; First posted 2019-10-25 (Actual); Results first posted 2024-02-08 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: capmatinib; pembrolizumab; NSCLC; PD-L1; EGFR; ALK; MET,; squamous; non-squamous
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — capmatinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Capmatinib 400mg BID + pembrolizumab 200mg Q3W (Experimental): Capmatinib (INC280) 400 mg orally twice daily (BID) in combination with pembrolizumab 200 mg intravenously every 3 weeks (Q3W)
  Interventions: Drug: Capmatinib; Biological: Pembrolizumab
- Pembrolizumab 200mg Q3W (Active Comparator): Pembrolizumab 200 mg intravenously every 3 weeks (Q3W)
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Drug: Capmatinib — INC280 tablets were administered orally at 400 mg on a continuous twice daily (BID) dosing schedule, from Day 1 until Day 21 of each 21-day cycle.
  Other Names: INC280
  Arms: Capmatinib 400mg BID + pembrolizumab 200mg Q3W
Biological: Pembrolizumab — Pembrolizumab was administered by intravenous infusion at 200 mg once every 3 weeks (Q3W).
  Other Names: Keytruda®; MK-3475

SUMMARY:
The purpose was to evaluate the efficacy and safety of the combination of capmatinib with pembrolizumab compared to pembrolizumab alone as first-line treatment for subjects with locally advanced or metastatic NSCLC who have PD-L1 expression ≥ 50% and have no EGFR mutation or ALK rearrangement. Capmatinib has demonstrated immunomodulatory activities when combined with an anti-PD1 antibody in preclinical tumor models irrespective of MET dysregulation. The combination of capmatinib with checkpoint inhibitors has been established to be tolerable and could provide additional clinical benefit to the subjects.

DETAILED DESCRIPTION:
This was a randomized, open-label, multicenter, phase II study evaluating the efficacy and safety of capmatinib plus pembrolizumab in comparison to pembrolizumab alone as first line treatment for locally advanced or metastatic non-small cell lung cancer (NSCLC) with programmed cell death ligand-1 (PD-L1) expression ≥ 50%, mesenchymal epithelial transition (MET) unselected, epidermal growth factor receptor (EGFR) wild type and anaplastic lymphoma kinase (ALK) negative.

All eligible subjects were randomized to one of the treatment arms in a 2:1 (capmatinib plus pembrolizumab: pembrolizumab alone) ratio. Participants in both treatment arms were to receive up to 35 cycles (approximately 24 months) of study treatment. The study enrollment was halted on 21-Jan-2021 per sponsor's decision. The enrollment halt decision was based on lack of tolerability observed in the capmatinib plus pembrolizumab arm.

Immediately following the enrollment halt, the below procedural changes were performed:

* Capmatinib treatment was discontinued in subjects on the combination arm. All ongoing subjects were allowed to continue receiving pembrolizumab single agent treatment as per investigator's discretion until unacceptable toxicity, or disease progression, or up to 35 cycles of treatment, whichever occurred first.
* Termination of capmatinib pharmacokinetics (PK) sample collection.
* Termination of pembrolizumab PK/immunogenicity (IG) sample collection. After the enrollment halt, the study protocol was amended (amendment 03) and the collection of efficacy data was stopped. As pembrolizumab is a registered and commercialized treatment for the study indication, the efficacy and safety assessments were to be performed as per each institution's standard of care and no longer captured in the electronic Case Report Form (eCRF) (except reporting of adverse events). Additionally, as single-agent pembrolizumab is a well-established standard treatment for the study indication, the requirement for post-treatment disease progression follow-up and survival follow-up were removed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed and documented locally advanced stage III (not candidates for surgical resection or definitive chemo-radiation) or stage IV (metastatic) NSCLC (per AJCC/IASLC v.8) for treatment in the first-line setting
* Histologically or cytologically confirmed diagnosis of NSCLC that is both EGFR wild type status and ALK- negative rearrangement statu
* Have an archival tumor sample or newly obtained tumor biopsy with high PD-L1 expression (TPS ≥ 50%)
* ECOG performance status score ≤ 1
* Have at least 1 measurable lesion by RECIST 1.1
* Have adequate organ function

Exclusion Criteria:

* Prior treatment with a MET inhibitor or HGF-targeting therapy
* Prior immunotherapy (e.g. anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways)
* Have untreated symptomatic central nervous system (CNS) metastases
* Clinically significant, uncontrolled heart diseases
* Prior palliative radiotherapy for bone lesions ≤ 2 weeks prior to starting study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2023-02-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- Australia (3):
  - Novartis Investigative Site, Wollongong, New South Wales
  - Novartis Investigative Site, North Adelaide, South Australia
  - Novartis Investigative Site, Shepparton, Victoria
- Novartis Investigative Site, Yvoir, Belgium
- Novartis Investigative Site, Québec, Quebec, Canada
- Novartis Investigative Site, Ostrava Vitkovice, Czechia
- France (3):
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
- Greece (2):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Thessaloniki
- Novartis Investigative Site, Shatin New Territories, Hong Kong, Hong Kong
- India (3):
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Kolkata, West Bengal
  - Novartis Investigative Site, Delhi
- Italy (2):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Aviano, PN
- Japan (2):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Yokohama, Kanagawa
- Malaysia (2):
  - Novartis Investigative Site, Kuching, Sarawak
  - Novartis Investigative Site, Kuala Lumpur
- Netherlands (3):
  - Novartis Investigative Site, Amersfoort
  - Novartis Investigative Site, Breda
  - Novartis Investigative Site, Zwolle
- Spain (5):
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Taiwan (2):
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Taichung
- Novartis Investigative Site, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2077

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 36 investigative sites in 16 countries.
Pre-assignment Details: The screening period began once patients had signed the study informed consent. Screening evaluations were performed within 28 days prior to the first dose of study treatment. After screening, the treatment period started on Cycle 1 Day 1.
Period: Overall Study
Arm/Group | Capmatinib 400mg BID + Pembrolizumab 200mg Q3W | Pembrolizumab 200mg Q3W
Started | 51 | 25
Entered Post-treatment Follow-up (Post-treatment disease progression follow-up and survival follow-up started on day 31 after last dose of study treatment. This was applicable until the implementation of Protocol Amendment 03.) | 38 | 20
Completed | 10 | 7
Not Completed | 41 | 18
Not completed — Adverse Event | 10 | 2
Not completed — Death | 6 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 3 | 1
Not completed — Progressive Disease | 19 | 9
Not completed — Subject Decision | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Capmatinib 400mg BID + Pembrolizumab 200mg Q3W | Pembrolizumab 200mg Q3W | Total
Number analyzed (Participants) | 51 | 25 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (7.59) | 66.6 (8.80) | 65.4 (8.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 9 | 25
  Male | 35 | 16 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 25 | 16 | 41
  Asian | 22 | 8 | 30
  Unknown | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) by Investigator Assessment as Per RECIST 1.1
Description: PFS is defined as the time from the date of randomization to the date of the first documented progression or death due to any cause. Tumor response was based on investigator assessment per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1.
  If a patient did not have an event, PFS was censored at the date of the last adequate tumor assessment, the start of a subsequent anti-neoplastic therapy (if any) or the date of sponsor's decision to discontinue capmatinib (applicable only to subjects on the combination arm).
  Due to the discontinuation of one of the investigational drugs (capmatinib) in all subjects in the combination arm, PFS was censored on the 21-Jan-2021 or the last adequate tumor assessment prior to that date for the capmatinib plus pembrolizumab arm.
  PFS was analyzed using Kaplan-Meier estimates.
Time Frame: Up to 1.3 years
Population: All patients to whom study treatment had been assigned by randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capmatinib 400mg BID + Pembrolizumab 200mg Q3W | Pembrolizumab 200mg Q3W
Number analyzed (Participants) | 51 | 25
months | 5.2 [2.0 to NA] — Not estimable due to insufficient number of participants with events. | 5.1 [2.6 to NA] — Not estimable due to insufficient number of participants with events.

2. Secondary Outcome: Overall Response Rate (ORR) by Investigator Assessment as Per RECIST 1.1
Description: Tumor response was based on local investigator assessment as RECIST v1.1. ORR per RECIST v1.1 is defined as the percentage of participants with a best overall response (BOR) of Complete Response (CR) or Partial Response (PR). For the capmatinib plus pembrolizumab arm, 21-Jan-2021 or any last adequate tumor assessment prior to that date was considered as the end of evaluation period for BOR.
  For RECIST v1.1, CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to 1.3 years
Population: All patients to whom study treatment had been assigned by randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Capmatinib 400mg BID + Pembrolizumab 200mg Q3W | Pembrolizumab 200mg Q3W
Number analyzed (Participants) | 51 | 25
Percentage of participants | 9.8 [3.3 to 21.4] | 40.0 [21.1 to 61.3]

3. Secondary Outcome: Disease Control Rate (DCR) by Investigator Assessment as Per RECIST 1.1
Description: Tumor response was based on local investigator assessment per RECIST v1.1. DCR is defined as the percentage of participants with a BOR of Complete Response (CR), Partial Response (PR), Stable Disease (SD), and non-CR/non-progressive disease (for subjects without target lesions). For the capmatinib plus pembrolizumab arm, 21-Jan-2021 or any last adequate tumor assessment prior to that date was considered as the end of evaluation period for BOR.
  For RECIST v1.1, CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters; SD= Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progression).
Time Frame: Up to 1.3 years
Population: All patients to whom study treatment had been assigned by randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Capmatinib 400mg BID + Pembrolizumab 200mg Q3W | Pembrolizumab 200mg Q3W
Number analyzed (Participants) | 51 | 25
percentage of participants | 37.3 [24.1 to 51.9] | 60.0 [38.7 to 78.9]

4. Secondary Outcome: Time to Response (TTR) by Investigator Assessment as Per RECIST 1.1
Description: TTR is defined as the time from the date of randomization to the first documented response of either complete response or partial response, which must be subsequently confirmed (although initial date of response is used, not date of confirmation).
  TTR was analyzed using the Kaplan-Meier method as defined in the statistical analysis plan.
Time Frame: Up to 1.3 years
Population: All patients to whom study treatment had been assigned by randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capmatinib 400mg BID + Pembrolizumab 200mg Q3W | Pembrolizumab 200mg Q3W
Number analyzed (Participants) | 51 | 25
months | NA [NA to NA] — Not estimable due to insufficient number of participants with events. | NA [NA to NA] — Not estimable due to insufficient number of participants with events.

5. Secondary Outcome: Duration of Response (DOR) by Investigator Assessment as Per RECIST 1.1
Description: DOR only applies to patients for whom best overall response is complete response (CR) or partial response (PR) based on local investigator assessment of overall lesion response according to RECIST v1.1. DOR is defined as the time from the date of first documented response (confirmed CR or confirmed PR) to the date of first documented disease progression or death due to any cause. If a patient not had an event, duration was censored at the date of last adequate tumor assessment before the start of a new anticancer therapy, if any.
  DOR was analyzed using the Kaplan-Meier method as defined in the statistical analysis plan.
Time Frame: Up to 1.3 years
Population: All patients to whom study treatment had been assigned by randomization and for whom best overall response was CR or PR as per RECIST v1.1 based on local investigator assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capmatinib 400mg BID + Pembrolizumab 200mg Q3W | Pembrolizumab 200mg Q3W
Number analyzed (Participants) | 5 | 10
months | NA [NA to NA] — Not estimable due to insufficient number of participants with events. | NA [NA to NA] — Not estimable due to insufficient number of participants with events.

6. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of randomization to the date of death due to any cause.
  The requirement for survival follow-up period was removed following the discontinuation of one of the investigational drugs (capmatinib) in all subjects in the combination arm and the implementation of Protocol Amendment 03.
  OS was analyzed using the Kaplan-Meier method as defined in the statistical analysis plan.
Time Frame: Up to 2.1 years
Population: All patients to whom study treatment had been assigned by randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capmatinib 400mg BID + Pembrolizumab 200mg Q3W | Pembrolizumab 200mg Q3W
Number analyzed (Participants) | 51 | 25
months | NA [NA to NA] — Not estimable due to insufficient number of participants with events. | NA [NA to NA] — Not estimable due to insufficient number of participants with events.

7. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Number of participants with AEs (any AE regardless of seriousness) and SAEs, including changes from baseline in vital signs, electrocardiograms and laboratory results qualifying and reported as AEs.
Time Frame: From first dose of study treatment to 30 days after last dose, up to 2.1 years
Population: All patients to whom study treatment had been assigned by randomization. Patients are analyzed according to the treatment they were randomized to.
Measure: Count of Participants; unit: Participants
Arm/Group | Capmatinib 400mg BID + Pembrolizumab 200mg Q3W | Pembrolizumab 200mg Q3W
Number analyzed (Participants) | 51 | 25
Participants
  AEs | 49 | 25
  Treatment-related AEs | 45 | 18
  SAEs | 31 | 13
  Treatment-related SAEs | 18 | 1
  AEs leading to discontinuation | 18 | 5
  Treatment-related AEs leading to discontinuation | 17 | 2
  AEs leading to dose reduction/interruption | 34 | 7
  Treatment-related AEs leading to dose reduction/interruption | 24 | 2

8. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Capmatinib
Description: Pharmacokinetic (PK) parameters were calculated based on capmatinib plasma concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed plasma concentration following a dose.
Time Frame: pre-dose and 1, 2, 4 and 8 hours after morning dose on Cycle 2 Day 1. The duration of one cycle was 21 days.
Population: Patients in the capmatinib pharmacokinetic analysis set (INC-PAS) with an available value for the outcome measure. INC-PAS consists of all patients who provided at least one blood sample with measurable capmatinib PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Capmatinib 400mg BID + Pembrolizumab 200mg Q3W
Number analyzed (Participants) | 25
ng/mL | 2730 (155.9)

9. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Capmatinib
Description: PK parameters were calculated based on capmatinib plasma concentrations by using non-compartmental methods. Tmax is defined as the time to reach maximum (peak) plasma concentration following a dose. Actual recorded sampling times were considered for the calculations.
Time Frame: pre-dose and 1, 2, 4 and 8 hours after morning dose on Cycle 2 Day 1. The duration of one cycle was 21 days.
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Arm/Group | Capmatinib 400mg BID + Pembrolizumab 200mg Q3W
Number analyzed (Participants) | 25
hours | 1.33 [0 to 4.00]

10. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of Capmatinib
Description: PK parameters were calculated based on capmatinib plasma concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUClast calculation.
Time Frame: pre-dose and 1, 2, 4 and 8 hours after morning dose on Cycle 2 Day 1. The duration of one cycle was 21 days.
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Capmatinib 400mg BID + Pembrolizumab 200mg Q3W
Number analyzed (Participants) | 25
hr*ng/mL | 4210 (232.8)

11. Secondary Outcome: Trough Serum Concentration (Ctrough) of Pembrolizumab
Description: PK parameters were calculated based on pembrolizumab serum concentrations by using non-compartmental methods. Ctrough is defined as the concentration reached immediately before the next dose is administered. All drug concentrations below the lower limit of quantification were treated as zero for the calculation of PK parameters.
Time Frame: pre-dose on Cycle 2 Day 1, Cycle 3 Day 1, Cycle 6 Day 1 and Cycle 12 Day 1. The duration of one cycle was 21 days.
Population: Patients in the pembrolizumab pharmacokinetic analysis set (Pembro-PAS) with an available value for the outcome measure at each timepoint. Pembro-PAS consists of all patients who provided at least one blood sample with measurable pembrolizumab PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Capmatinib 400mg BID + Pembrolizumab 200mg Q3W | Pembrolizumab 200mg Q3W
Number analyzed (Participants) | 32 | 18
µg/mL
  Cycle 2 Day 1 | 11.8 (37.5) | 10.6 (34.8)
  Cycle 3 Day 1: number analyzed (Participants) | 29 | 18
  Cycle 3 Day 1 | 18.9 (51.9) | 18.2 (32.3)
  Cycle 6 Day 1: number analyzed (Participants) | 14 | 8
  Cycle 6 Day 1 | 27.6 (66.5) | 36.8 (26.0)
  Cycle 12 Day 1: number analyzed (Participants) | 0 | 2
  Cycle 12 Day 1 |  | 49.7 (10.0)

12. Secondary Outcome: Number of Participants With Anti-pembrolizumab Antibodies
Description: Immunogenicity (IG) was evaluated in serum samples. The assay to quantify and assess the IG was a validated homogeneous enzyme-linked immunosorbent assay (ELISA).
  * ADA-negative at baseline: ADA-negative sample at baseline
  * ADA-positive at baseline: ADA-positive sample at baseline
  * ADA-negative post-baseline: patient with ADA-negative sample at baseline and at least 1 post baseline determinant sample, all of which are ADA-negative samples
  * ADA-positive post-baseline: patient with at least 1 ADA-positive sample post baseline
Time Frame: Baseline (pre-dose), up to 8 months
Population: All patients to whom study treatment had been assigned by randomization and who had a determinant baseline IG sample and at least one determinant post-baseline IG sample. A determinant sample is neither ADA-inconclusive nor unevaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Capmatinib 400mg BID + Pembrolizumab 200mg Q3W | Pembrolizumab 200mg Q3W
Number analyzed (Participants) | 42 | 20
Participants
  ADA-negative at baseline | 37 | 18
  ADA-positive at baseline | 5 | 2
  ADA-negative post-baseline | 36 | 18
  ADA-positive post-baseline | 6 | 2

13. Post Hoc Outcome: All-Collected Deaths
Description: On-treatment deaths were collected from start of treatment to 30 days after last dose.
  Post-treatment survival follow-up deaths were collected from day 31 after last dose of study treatment until the requirement for survival follow-up was removed following the discontinuation of capmatinib in the combination arm (protocol amendment 03).
  All deaths refer to the sum of on-treatment deaths plus post-treatment survival follow-up deaths.
Time Frame: On-treatment: Up to 2.1 years after start of treatment. Post-treatment survival follow-up: Up to 1.3 years after start of treatment.
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Capmatinib 400mg BID + Pembrolizumab 200mg Q3W | Pembrolizumab 200mg Q3W
Number analyzed (Participants) | 51 | 25
participants
  On-treatment deaths | 10 | 3
  Post-treatment survival follow-up deaths: number analyzed (Participants) | 38 | 20
  Post-treatment survival follow-up deaths | 6 | 5
  All deaths | 16 | 8

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment to 30 days after last dose, up to 2.1 years after start of treatment. Deaths were collected in the post-treatment survival follow-up from day 31 after last dose of study treatment until the requirement for survival follow-up was removed following the discontinuation of capmatinib in the combination arm (protocol amendment 03), up to 1.3 years after start of treatment. These are not considered AEs.
Description: Patients were analyzed according to the treatment they actually received. Deaths in the post-treatment survival follow-up are not considered Adverse Events. The total number at risk in the post treatment survival includes patients that entered the post treatment survival follow-up period.
Groups:
- Capmatinib + Pembrolizumab - On-treatment: Capmatinib 400 mg BID in combination with pembrolizumab 200 mg Q3W. AEs collected during on-treatment period (up to 30 days after last dose).
- Pembrolizumab After Combination Treatment - On-treatment: Pembrolizumab single agent 200 mg Q3W after discontinuing capmatinib. AEs collected during on-treatment period (up to 30 days after last dose).
- Pembrolizumab - On-treatment: Pembrolizumab single agent 200 mg Q3W from study start. AEs collected during on-treatment period (up to 30 days after last dose).
- Capmatinib + Pembrolizumab - Post-treatment Survival Follow-up: Capmatinib 400 mg BID in combination with pembrolizumab 200 mg Q3W. Deaths collected in the post-treatment follow-up period (starting from day 31 after last dose). No AEs were collected during this period.
- Pembrolizumab - Post-treatment Survival Follow-up: Pembrolizumab single agent 200 mg Q3W from study start. Deaths collected in the post-treatment follow-up period (starting from day 31 after last dose). No AEs were collected during this period.
Arm/Group | Capmatinib + Pembrolizumab - On-treatment | Pembrolizumab After Combination Treatment - On-treatment | Pembrolizumab - On-treatment | Capmatinib + Pembrolizumab - Post-treatment Survival Follow-up | Pembrolizumab - Post-treatment Survival Follow-up
All-Cause Mortality (participants affected / at risk) | 8/51 | 2/51 | 3/25 | 6/38 | 5/20
Serious Adverse Events (participants affected / at risk) | 26/51 | 9/51 | 13/25 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 41/51 | 29/51 | 24/25 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Capmatinib + Pembrolizumab - On-treatment (N=51) | Pembrolizumab After Combination Treatment - On-treatment (N=51) | Pembrolizumab - On-treatment (N=25) | Capmatinib + Pembrolizumab - Post-treatment Survival Follow-up (N=0) | Pembrolizumab - Post-treatment Survival Follow-up (N=0)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | NA | NA
Cardiac failure (Cardiac disorders) | 1 | 0 | 1 | NA | NA
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | NA | NA
Pericardial effusion (Cardiac disorders) | 1 | 2 | 0 | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA
Disease progression (General disorders) | 1 | 0 | 0 | NA | NA
General physical health deterioration (General disorders) | 1 | 0 | 1 | NA | NA
Pyrexia (General disorders) | 3 | 1 | 0 | NA | NA
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0 | NA | NA
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 0 | NA | NA
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | NA | NA
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | NA | NA
Bronchitis (Infections and infestations) | 2 | 0 | 1 | NA | NA
Cellulitis (Infections and infestations) | 0 | 1 | 0 | NA | NA
Encephalitis (Infections and infestations) | 1 | 0 | 0 | NA | NA
Meningitis listeria (Infections and infestations) | 1 | 0 | 0 | NA | NA
Myelitis (Infections and infestations) | 0 | 0 | 1 | NA | NA
Pneumonia (Infections and infestations) | 2 | 1 | 2 | NA | NA
Sepsis (Infections and infestations) | 2 | 1 | 0 | NA | NA
Septic shock (Infections and infestations) | 1 | 0 | 0 | NA | NA
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA
Transaminases increased (Investigations) | 1 | 0 | 0 | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | NA | NA
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | NA | NA
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | NA | NA
Brain oedema (Nervous system disorders) | 1 | 0 | 0 | NA | NA
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | NA | NA
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0 | NA | NA
Seizure (Nervous system disorders) | 1 | 0 | 0 | NA | NA
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 0 | NA | NA
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | NA
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | NA
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | NA
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | NA | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | NA
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | NA | NA
Hypotension (Vascular disorders) | 1 | 0 | 0 | NA | NA
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1 | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Capmatinib + Pembrolizumab - On-treatment (N=51) | Pembrolizumab After Combination Treatment - On-treatment (N=51) | Pembrolizumab - On-treatment (N=25) | Capmatinib + Pembrolizumab - Post-treatment Survival Follow-up (N=0) | Pembrolizumab - Post-treatment Survival Follow-up (N=0)
Anaemia (Blood and lymphatic system disorders) | 4 | 2 | 0 | NA | NA
Tachycardia (Cardiac disorders) | 0 | 0 | 2 | NA | NA
Hypothyroidism (Endocrine disorders) | 1 | 6 | 1 | NA | NA
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2 | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 3 | 3 | 1 | NA | NA
Constipation (Gastrointestinal disorders) | 5 | 7 | 4 | NA | NA
Diarrhoea (Gastrointestinal disorders) | 8 | 4 | 6 | NA | NA
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 2 | NA | NA
Nausea (Gastrointestinal disorders) | 13 | 1 | 2 | NA | NA
Vomiting (Gastrointestinal disorders) | 14 | 1 | 2 | NA | NA
Asthenia (General disorders) | 4 | 1 | 5 | NA | NA
Chest pain (General disorders) | 2 | 2 | 3 | NA | NA
Chills (General disorders) | 3 | 0 | 0 | NA | NA
Fatigue (General disorders) | 2 | 3 | 5 | NA | NA
Oedema peripheral (General disorders) | 14 | 6 | 1 | NA | NA
Pyrexia (General disorders) | 9 | 2 | 5 | NA | NA
Hypersensitivity (Immune system disorders) | 0 | 1 | 2 | NA | NA
COVID-19 (Infections and infestations) | 0 | 0 | 2 | NA | NA
Alanine aminotransferase increased (Investigations) | 11 | 4 | 3 | NA | NA
Amylase increased (Investigations) | 4 | 3 | 2 | NA | NA
Aspartate aminotransferase increased (Investigations) | 11 | 2 | 3 | NA | NA
Blood alkaline phosphatase increased (Investigations) | 5 | 0 | 1 | NA | NA
Blood bilirubin increased (Investigations) | 6 | 1 | 1 | NA | NA
Blood creatine phosphokinase increased (Investigations) | 1 | 3 | 0 | NA | NA
Blood creatinine increased (Investigations) | 7 | 1 | 1 | NA | NA
Blood lactate dehydrogenase increased (Investigations) | 3 | 1 | 0 | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 4 | 0 | 2 | NA | NA
Lipase increased (Investigations) | 2 | 2 | 2 | NA | NA
SARS-CoV-2 test negative (Investigations) | 4 | 0 | 2 | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 5 | 2 | 5 | NA | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 | 2 | 2 | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 3 | 0 | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 5 | 6 | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 3 | NA | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3 | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | NA | NA
Dizziness (Nervous system disorders) | 1 | 1 | 3 | NA | NA
Headache (Nervous system disorders) | 3 | 1 | 3 | NA | NA
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 3 | NA | NA
Paraesthesia (Nervous system disorders) | 1 | 1 | 4 | NA | NA
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 2 | NA | NA
Insomnia (Psychiatric disorders) | 4 | 3 | 4 | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 4 | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 3 | NA | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | NA | NA
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | NA | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | NA | NA
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | NA | NA
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | NA | NA
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 7 | 8 | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 5 | 5 | 3 | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | NA | NA
Hypertension (Vascular disorders) | 1 | 0 | 6 | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT04139317/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT04139317/SAP_001.pdf